CLINICAL TRIAL: NCT01378936
Title: Phase 2 RCT of Jail-Based Impact of Crime Intervention to Reduce Recidivism, Substance Abuse and HIV Risk Behavior
Brief Title: Jail-Based Impact of Crime Intervention
Acronym: IOC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: George Mason University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, June Tangney, Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA014694-11 (NIH); R01DA014694 (NIH)
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Substance Abuse; HIV Risk; Criminogenic Thinking; Shame; Guilt; Empathy
Keywords: criminal behavior; substance abuse; HIV risk behavior; criminogenic thinking; shame; guilt; empathy; jail inmates; restorative justice; crime
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MI plus IOC group intervention (Experimental)
  Interventions: Behavioral: MI plus IOC group intervention
- Motivational Interview only (Experimental)
  Interventions: Behavioral: Motivational Interview only

INTERVENTIONS:
Behavioral: MI plus IOC group intervention — 45 minute Motivational Interview plus 16 session IOC intervention
  Other Names: Impact of Crime
  Arms: MI plus IOC group intervention
Behavioral: Motivational Interview only — 45 minute Motivational Interview session
  Arms: Motivational Interview only

SUMMARY:
The purpose of this study is to evaluate whether the Impact of Crime (IOC) group intervention with jail inmates reduces post-release recidivism, substance abuse, and HIV risk behavior.

DETAILED DESCRIPTION:
This project imports social-personality theory and research on moral emotions and cognitions to the applied problems of crime, substance abuse, and HIV risk behavior. The primary aim of this study, a Phase 2 Randomized Clinical Trial (RCT) of the restorative justice-inspired Impact of Crime (IOC) group intervention, is to examine the efficacy of treatment and to determine if changes in moral emotions and cognitions serve as mechanisms of action, explaining the impact of treatment involvement on reductions in post-release recidivism, substance abuse, and HIV risk behavior.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must be male
* Must be currently incarcerated jail inmate
* Must be sentenced
* Sentence must be short enough to serve out sentence at ADC
* Release date must follow projected final session of treatment
* Must speak, read, and write in English with sufficient proficiency to use workbook and participate in group sessions
* Must be assigned to the jail's "general population"

Exclusion Criteria:

* Actively psychotic
* Assigned "keep separate" from other group members

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Recidivism - Self report of arrests and undetected crimes | 3 months post-release
Recidivism - Self report of arrests and undetected crimes | 1 yr post-release
Recidivism - Self report of arrests and undetected crimes | 3 yr post-release
Recidivism - Self report of arrests and undetected crimes | 5 yr post-release
Recidivism -- official FBI records of arrests | 1 yr post-release
Recidivism -- official FBI records of arrests | 3 yr post-release
Recidivism -- official FBI records of arrests | 5 yr post-release

SECONDARY OUTCOMES:
Changes in self-reported shame-proneness from baseline | changes from baseline to post tx and 3 mo, 1 yr, 3yr and 5 yr post-release
Changes in self-reported guilt proneness from baseline | changes from baseline to post tx, and 3 mo, 1 yr, 3 yr, 5 yr post-release
Changes from self-reported empathy from baseline | changes from baseline to post tx, 3 mo, 1 yr, 3 yr, 5 yr post-release
Changes from self-reported criminogenic thinking at baseline | changes from baseline to post tx, and 3 mo, 1 yr, 3 yr, 5 yr post-release
Changes in self-reported substance use and dependence from 1 yr pre-incarceration | changes from pre-incarceration to 3 mo, 1 yr, 3 yr, 5 yr post-release
Changes in self-reported HIV risk behavior (sex and IDU) from 1 year pre-incarceration | changes from pre-incarceration to 3 mo, 1 yr, 3 yr, 5 yr post-release

CONTACTS AND LOCATIONS:
Overall Officials: June P Tangney, Ph.D., Principal Investigator — George Mason University
Locations (1):
- Fairfax County Adult Detention Center, Fairfax, Virginia, United States